CLINICAL TRIAL: NCT01558596
Title: Cardiac Remote Ischemic Preconditioning Prior to Elective Major Vascular Surgery
Brief Title: Remote Ischemic Preconditioning Prior to Vascular Surgery
Acronym: CRIPES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLIN-014-11F
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Peripheral Arterial Disease; Vascular Surgery
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham (Placebo Comparator): Blood pressure cuff inflated to 40-50 mmHg in the upper extremity
  Interventions: Procedure: Control
- RIPC (Experimental): Blood pressure cuff inflated to 200 mmHg in the upper extremity for 5 minutes to cause forearm ischemia by external compression of the brachial artery. This will be followed by 5 minutes of cuff deflation to allow for preperfusion. The ischemia-reperfusion cycle will be repeated 3 times for a total duration of 30 minutes, equally divided between ischemia and reperfusion.
  Interventions: Procedure: Preconditioning

INTERVENTIONS:
Procedure: Preconditioning — Blood pressure cuff inflated to 200 mmHg in the upper extremity for 5 minutes to cause forearm ischemia by external compression of the brachial artery. This will be followed by 5 minutes of cuff deflation to allow for preperfusion. The ischemia-reperfusion cycle will be repeated 3 times for a total duration of 30 minutes, equally divided between ischemia and reperfusion.
  Arms: RIPC
Procedure: Control — Blood pressure cuff inflated to 40-50 mmHg in the upper extremity
  Arms: Sham

SUMMARY:
The investigators have previously shown that elective vascular surgery is a high-risk operation with an anticipated risk of either death or heart attack of 15%. This study is testing whether a protocol of remote ischemic preconditioning (RIPC) applied 24 hours prior to the operation is safe, feasible and reduces the incidence of an adverse, perioperative cardiac complication.

DETAILED DESCRIPTION:
The proposed investigation has a single blind, randomized design and plans to enroll 180-205 patients who are scheduled to have major, elective vascular surgery for occlusive carotid disease, expanding abdominal aortic aneurysm (AAA), occlusive lower extremity disease and/or critical limb ischemia at the Minneapolis VA Health Care Center. 24 hours prior to the patient's scheduled vascular operation, RIPC therapy will be applied to one of the participant's upper arms to cause forearm ischemia. Clinically collected, pre-operative troponins, creatine kinase MBs (CK-MBs), EKGs along with troponins, CK-MBs and EKGs collected on day 1, 2, 3 and day 7 (if still hospitalized) will be utilized to evaluate the occurrence of perioperative, adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective major vascular surgery at the Minneapolis VA Medical Center for abdominal aortic aneurysm, carotid disease or limb ischemia.
* Age > 18.
* Provides informed consent.

Exclusion Criteria:

* Hypertensive crisis
* Peripheral arterial disease of the upper extremities
* Arteriovenous (AV) fistula
* Acute Coronary Syndrome (ACS) in the last 6 months
* Severe valvular heart disease
* Pregnant women
* Unable to provide consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santiago A Garcia, MD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garcia S, Rector TS, Zakharova M, Herrmann RR, Adabag S, Bertog S, Sandoval Y, Santilli S, Brilakis ES, McFalls EO. Cardiac Remote Ischemic Preconditioning Prior to Elective Vascular Surgery (CRIPES): A Prospective, Randomized, Sham-Controlled Phase II Clinical Trial. J Am Heart Assoc. 2016 Sep 29;5(10):e003916. doi: 10.1161/JAHA.116.003916. PMID 27688236
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: From June 2011 to September 2015
Pre-assignment Details: A total of 205 patients were randomized, of which 201 received treatment. 4 patients removed from study after randomization
Period: Overall Study
Arm/Group | Sham | RIPC
Started | 104 | 101
Completed | 101 | 100
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — surgery elsewhere or cancelled | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | RIPC | Total
Number analyzed (Participants) | 101 | 100 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (7) | 69 (7) | 69 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 101 | 100 | 201
Region of Enrollment [Number; unit: participants]
  United States | 101 | 100 | 201

OUTCOME MEASURES:

1. Primary Outcome: Troponin I Elevation Above the Upper Reference Limit (URL)
Description: Troponin I is a biomarker of myocardial necrosis that may indicate myocardial damage or injury that occurs during the perioperative period
Time Frame: Within 3 days of the vascular operation
Measure: Number; unit: participants
Groups:
- Sham: Blood pressure cuff inflated to 40-50 mmHg over brachial artery
- RIPC: Blood pressure cuff inflated to 200 mmHg over the brachial artery while confirming absence of radial and ulnar pulse. Total duration of protocol was 30 minutes, equally divided between reperfusion and ischemia.
Arm/Group | Sham | RIPC
Number analyzed (Participants) | 101 | 100
participants | 25 | 22

ADVERSE EVENTS:
Groups:
- Sham: Blood pressure cuff inflated to 40 mmHg to mask controls
- RIPC: Blood pressure cuff inflated above systolic blood pressure (200 mmHg) over brachial artery to induce forearm ischemia. Total duration of protocol 30 minutes equally divided between ischemia ( 5 minutes x 3) and reperfusion ( 5 minutes x3)
Arm/Group | Sham | RIPC
Serious Adverse Events (participants affected / at risk) | 8/101 | 5/100
Other Adverse Events (participants affected / at risk) | 0/101 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=101) | RIPC (N=100)
Myocardial infarction (Cardiac disorders) | 1 (2) | 1 (1)
Cellulitis (Surgical and medical procedures) | 5 (5) | 3 (3) — Cellulitis/surgical site infection
Stroke (Cardiac disorders) | 1 (1) | 0 (0)
heart failure (Cardiac disorders) | 0 (0) | 1 (1)
pacemaker (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes